CLINICAL TRIAL: NCT06100185
Title: Wearable Neurotechnology for Treatment of Insomnia (tES)
Brief Title: Wearable Transcranial Electrical Stimulation (tES) for Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: WNTI-2022
Record Dates: First submitted 2023-07-28; First posted 2023-10-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-06

CONDITIONS: Insomnia
Keywords: tES; Insomnia; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Experimental Arm (Experimental)
  Interventions: Device: PeakSleep
- Sham Arm (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: PeakSleep — The PeakSleepTM is a constant current device which delivers stable stimulation as a function of the impedance measured across the electrodes (e.g. it varies voltage to produce a steady current). The device gradually ramps up the current as the impedance decreases during the stimulation session. The device uses stimulation amplitudes in the range of 100uA to 500uA at each electrode pair. Devices will be configured to deliver 100 stimulation trains over 30 minutes where each train is 6 pulses of 0.75Hz trapezoidal stimulation (each train lasts 8 seconds). The inter-train interval is 10 seconds leading to a total stimulation time of <14 minutes with a maximum dose of 1mA (500uA per electrode pair).
  Arms: Experimental Arm
Device: Sham — Sham is delivered with the same devices which are alternatively configured to deliver a trivially low amplitude (e.g. 100uA) waveform of a different frequency (e.g. 25 Hz) for the same treatment duration. Beyond differences in amplitude and frequency of stimulation, devices will be operated in exactly the same way during sham treatment.
  Arms: Sham Arm

SUMMARY:
The purpose of this study is to investigate the ability of a translational device, Teledyne PeakSleep, to reduce sleep onset latency, reduce time awake after sleep onset and improve restfulness and the subjective benefits of sleep in a patient population with insomnia via transcranial direct current stimulation (tDCS) applied to frontal lobe circuits.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate a new, targeted intervention to improve outcomes for those suffering from insomnia by attempting to enhance the brain rhythms within the frontal lobe implicated in slow wave generation during the transition from wake to sleep. The device applies a pulsed trapezoidal direct current waveform at 0.75 Hz to the frontal areas of the brain immediately prior to attempted sleep onset to facilitate the transition to sleep.

During this cross-over trial, patients will be asked to use a PeakSleep wearable neurotechnology prototype headband, which delivers <14 minutes of frontal tDCS over a 30-minute period, immediately before trying to fall asleep. Using an active stimulation versus sham paradigm, we will compare actigraphy data, physiological data, and subjective sleep measures against a pre-treatment baseline in the same patient.

Participants will complete five in-person visits over the course of the 8-week study. The first visit includes the collection of baseline self-reported data and actigraphy device training. All subsequent visits involve headset training, downloading PeakSleep and actigraphy data, repeating self-reported data measures, and reporting user experience with the device. Participants will not perform any formal sleep study visits and instead provide daily actigraphy data via a FitBit and EEG data when wearing PeakSleep in their own home.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with sleep onset insomnia
* Self report insomnia diagnosis (ISI score ≥15)
* 18-70 years old that are Tricare eligible
* No pharmacologic or non-pharmacologic treatment for insomnia in the last 14 days, including over-the-counter medications such as diphenhydramine or cyclobenzaprine not using sedating medications (including over-the-counter) at bedtime in the last 14 days. These can include sedating antihistamines such as diphenhydramine/Benadryl, combination pills such as Tylenol or Advil PM, ZzzQuil. Psychiatric medications such as benzodiazepines (clonazepam/Klonopin, lorazepam/Ativan, diazepam/Valium, alprazolam/Xanax), anti-histamines (hydroxyzine/Atarax/Vistaril), or anti-psychotics (quetiapine/Seroquel).

Exclusion Criteria:

* Neurologic conditions such as seizures or conditions that increase the risk of seizures, including concussions within the last 3 months; moderate or severe traumatic brain injury; stroke; multiple sclerosis; or cognitive impairment with or without the use of prescription medication or requirement for hospitalization.
* Any psychiatric disorder requiring weekly or more frequent clinical monitoring or medication changes in the last 4 weeks.
* History of neurodevelopmental disorder such as attention deficit hyperactivity disorder, learning disability, or developmental delay
* Any inpatient hospitalization, major surgery, or medical procedure within the past 6 months
* Hearing impairments requiring implanted or external devices worn at all times for amplification.

  **Pregnant or believes there is a chance of pregnancy
* Current substance use disorder (addiction) within the past year, not including nicotine Current use of narcotics (opioid based medications for the treatment of pain (OxyContin, Percocet, Vicodin, etc.) with or without a prescription within the last year
* Change in psychotropic (non sleep related) medications within the last 4 weeks (examples include: benzodiazepines, SSRI/SNRIs, bupropion, gabapentin).
* Consuming more than 10 alcoholic beverages per week
* Treatment for drug or alcohol use/abuse within the past 1 year
* Presence of a recently diagnosed or unstable sleep disorder, other than insomnia, with an treatment regimen less than 3 months old
* Any motor coordination deficits that interfere with use of the tES device
* Participants should not have trauma/cuts/rashes to their forehead or behind the ears that would interfere with wearing of the device or cause discomfort for the research subject
* Tattoos on the head
* Non-removable metal above the shoulders, except bridges or fillings, OR implanted devices anywhere in the body (e.g., pacemakers, defibrillators, cochlear implants, brain implants including deep brain stimulators or other implanted devices) presence of an unstable medical condition that significantly contributes to their insomnia (e.g. chronic pain, cough, GERD, sleep apnea) - or diagnosis of an above condition that no longer significantly contribute to insomnia but has not been stable on a treatment regimen for at least 3 months.

any suicidal attempts within the last 12 months.

* Any other condition that the investigator believes would prevent completion of the study or put participant at risk
* Any suicidal ideations or thoughts of self-harm (as measured by the PHQ-9, Item 9) within the last 2 weeks.

  * Note: Pregnancy Safety data for tES use in pregnant women is scarce but is reviewed in: Antal, Andrea, et al. "Low intensity transcranial electric stimulation: safety, ethical, legal regulatory and application guidelines." Clinical neurophysiology 128.9 (2017): 1774-1809. The authors cite two case studies of tES use in pregnant women with no impact or safety risk for the mother or fetus when tES was applied to the head at 2mA and 20-30 min per day. The recommendation by the authors is to verbally enquire as to the pregnancy status of the subjects and only deliver tES when the benefit outweighs risk. Here we propose to completely exclude this population if the questionnaire reveals they are pregnant or are trying to become pregnant. In the event that the patient is untruthful regarding their pregnancy status we view the risk as insignificant given these reported studies and the fact that our dose is <¼ the dose used in them. For this reason we have chosen not to perform a urine test to screen for pregnancy as we view it as an obtrusive and unnecessary step given the risk profile.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Onset Latency Change from Baseline | 5 weeks
  FitBit actigraphy data will be collected to measure daily sleep onset latency (SOL) for two weeks at baseline (weeks 1-2, averaged) and compared to that of the study period (weeks 3-5).

SECONDARY OUTCOMES:
ISI Change from Baseline | 5 weeks
  The Insomnia Severity Index (score from 0-28, higher is worse insomnia) will capture sleep habits and insomnia symptomatology during experimental sessions. Compared across pre-screen and 5 visit blocks.
PHQ-9 Change from Baseline | 5 weeks
  The Patient Health Questionnaire (PHQ-9, score from 0-27, higher is worse depression) will assess psychiatric conditions at visits 1, 3, and 5.
Total Sleep Time Change from Baseline | 5 weeks
  FitBit actigraphy data will be collected to measure total sleep time (TST) and time awake after sleep onset (WASO) during the first treatment block, for two weeks. During weeks 3-5.
EEG spectral changes from baseline (Delta power increase) | 5 weeks
  The PeakSleep device contains 3 EEG sensors (approximately Fp1, Fpz, Fp2) which will collect EEG data for investigation of neural activity for both stimulation and sham conditions. Will occur nightly for two weeks during Treatment 1 (i.e., weeks 3-4).
Heart rate variability change from baseline | 5 weeks
  For two weeks during treatment 1, heart rate will be collected daily via FitBit. Averages will be averages compared across treatment blocks (baseline, treatment 1, washout, treatment 2)

CONTACTS AND LOCATIONS:
Overall Officials: John K Werner, MD PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The specific individual participant data (IPD) to be shared includes de-identified EEG recordings collected during treatment sessions and responses to sleep diary questions. This data is coded using an alphanumeric identifier unlinked from any personal information. The mapping spreadsheet linking identifiers to participants will be destroyed 120 days after study completion, fully de-identifying the data. Participants consent to future use of their data through an opt-in checkbox and may withdraw consent at any time. Only approved research staff will access the data, stored securely per DoD and USUHS guidelines.
Supporting Information: Study Protocol
Time Frame: The de-identified individual participant data (IPD) and supporting information will be available starting 120 days after study completion, following destruction of the spreadsheet linking participant identities to study codes. The data will be maintained indefinitely by Dr. Werner for future research use, with no specified end date.
Access Criteria: Only research staff listed in the study protocol and approved by the IRB will have access to the IPD and supporting information. They will be able to access de-identified EEG data and sleep diary responses linked only to alphanumeric codes. Access will be through secure, password-protected computers or servers. After de-identification, the data may be shared for future research with qualified investigators upon request and IRB approval, but will remain free of any personal identifiers and only include data necessary for approved analyses.